CLINICAL TRIAL: NCT06593665
Title: Randomized Prospective Study Comparing Intrathecal Morphine Vs Intravenous Methadone for Postoperative Analgesia Following Retroperitoneal Lymph Node Dissection (RPLND)
Brief Title: Intrathecal Morphine Versus Intravenous Methadone for Postoperative Analgesia Following Retroperitoneal Lymph Node Dissection.
Acronym: RPLND
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Gulraj Chawla, Dept. of Anesthesiology, Asst. Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 22103
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 142 subjects will be randomized by a computer program into two groups.
  1. Intrathecal preservative free morphine (duramorph) 200mcg with 7.5 mg of hyperbaric bupivacaine placed by a spinal needle prior to induction of general anesthesia (n=71)
  2. Intravenous methadone dose at 0.2mg/kg Ideal Body weight up to a maximum dose of 20 mg, rounded to the nearest milligram, for all patients given during the induction of general anesthesia (n=71)
Who Masked: Participant, Care Provider
Masking Description: The primary investigator or his/her designee will inform the anesthesiology team caring for each subject of the arm of the study they are in for each case. Subjects and research staff doing post-operative assessments will be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Morphine (Other): Intrathecal preservative free morphine (duramorph) 200 mcg with 7.5mg of hyperbaric bupivacaine placed by a spinal needle prior to induction of general anesthesia (n=71)
  Interventions: Drug: Inrathecal Morphine
- Intravenous Methadone (Other): Intravenous methadone dosed at 0.2 mg/kg Ideal Body weight up to a maximum dose of 20mg, rounded to the nearest milligram, for all patients given during the induction of general anesthesia (n=71)
  Interventions: Drug: Intravenous Methadone

INTERVENTIONS:
Drug: Inrathecal Morphine — Intrathecal preservative free morphine (duramorph) 200 mcg with 7.5mg of hyperbaric bupivacaine placed by a spinal needle prior to induction of general anesthesia (n=71)
  Arms: Intrathecal Morphine
Drug: Intravenous Methadone — Intravenous methadone dosed at 0.2 mg/kg Ideal Body weight up to a maximum dose of 20mg, rounded to the nearest milligram, for all patients given during the induction of general anesthesia (n=71)
  Arms: Intravenous Methadone

SUMMARY:
This randomization study is to compare both intrathecal morphine and intravenous methadone, which are both standard of care, for pain management in patients undergoing retroperitoneal lymph node dissections for primary testicular cancer. Investigators plan to compare their analgesic effectiveness at different postoperative time intervals.

DETAILED DESCRIPTION:
In this study, investigators aim to compare intravenous methadone combined with standard multimodal analgesia and surgical infiltration of local anesthesia to intrathecal duramorph with standard multimodal analgesia and surgical infiltration of local anesthesia. In this single blinded prospective randomized control trial, investigators hypothesize that intravenous methadone will provide a significant reduction in patient opioid consumption when compared to intrathecal opioid analgesia in the first 24 hours in patients who undergo PC/RPLND.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a virgin (chemotherapy has not been used) or post- chemotherapy retroperitoneal lymph node dissection for primary testicular cancer at IU Health AAHC
* ASA Class 1, 2, 3
* Age 18 to 80 years; Male
* BMI less than 50kg/m2

Exclusion Criteria:

* Any contraindication for neuraxial analgesia
* Patient on home methadone at any dose
* Any physical, mental or medical conditions which, in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* Known true allergy to the study medications (morphine, bupivacaine, acetaminophen, methadone)
* Any history of substance abuse in the past 6 months which would include heroin or any other illegal street drugs
* End stage liver disease, end stage renal disease
* Patient staying intubated after surgery
* Patient (home dose) taking more than 30mg PO morphine equivalent (PME) per day
* Any additional surgical procedures to the patient with a different surgical incision compared to the standard laparotomy for the RPLND procedure, i.e. thoracic tumor reduction

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 142 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
IV morphine equivalent (MME) | First 24 hours postoperative
  Cumulative Milligrams of morphine equivalent (MME) consumption

SECONDARY OUTCOMES:
Opioid consumption | 1 hour after arrival time to post anesthesia care unit
  Opioid consumption in morphine equivalent (MME)
Opioid consumption | 12 hours after arrival time to post anesthesia care unit
  Opioid consumption in morphine equivalent (MME)
Opioid consumption | 24 hours after arrival time to post anesthesia care unit
  Opioid consumption in morphine equivalent (MME)
Opioid side effect-Nausea | after arrival time to post anesthesia care unit until 24 hours/completion of study
  Incidence of opioid side effects-nausea
Opioid side effects-Vomiting | after arrival time to post anesthesia care unit until 24 hours/completion of study
  Incidence of opioid side effects-vomiting
Opioid side effects-Pruritis | after arrival time to post anesthesia care unit until 24 hours/completion of study
  Incidence of opioid side effects-pruritis
Adverse Events | after arrival time to post anesthesia care unit until 24 hours/completion of study
  Incidence of adverse events
Opioid side effects-Respiratory Depression | after arrival time to post anesthesia care unit until 24 hours/completion of study
  Incidence of opioid side effects-respiratory depression
Pain Scores | 24 hours after arrival time to post anesthesia care unit
  Visual Analog Scale (VAS) pain score On a scale of 1 to 10 (increments of 1 unit), 1 being no pain at all, 10 being the most pain the patient has ever experienced
Pain Scores | 12 hours after arrival time to post anesthesia care unit
  Visual Analog Scale (VAS) pain score On a scale of 1 to 10 (increments of 1 unit), 1 being no pain at all, 10 being the most pain the patient has ever experienced

CONTACTS AND LOCATIONS:
Overall Officials: Gulraj S Chawla, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana Univeristy, Indianapolis, Indiana
  - Indiana University Hospital, Indianapolis, Indiana